CLINICAL TRIAL: NCT03149146
Title: Improving Clinical Decision Making Skills of Physical Therapists in Myanmar By Series of Educational Workshop
Brief Title: Improving Clinical Decision Making Skills for Myanmar Physical Therapists by Series of Workshop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: University of Medical Technology, Yangon (Other)
Responsible Party: Principal Investigator, PHYU HNIN HLAING, PhD candidate, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU
Record Dates: First submitted 2017-05-08; First posted 2017-05-11 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Cognitive Change
Keywords: Clinical Decision Making; Myanmar Physical therapists; Educational workshop

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Decision Making (CDM) Workshop (Experimental): Series of CDM educational workshop will be conducted for one group of participants and they will be guided the CDM process through the two clinical practice models; Therapeutic process (TP) and International Classification of Functioning, Disability and Health (ICF).
  Interventions: Other: Clinical Decision Making (CDM) Workshop
- Clinical Decision Making Workbook (Active Comparator): Participants will receive Clinical Decision Making (CDM) workbook which will be used to teach the Clinical Decision Making process in the four days workshop.
  Interventions: Other: Clinical Decision Making (CDM) Workbook

INTERVENTIONS:
Other: Clinical Decision Making (CDM) Workshop — Participants will be provided the Clinical Decision Making workbook which will be used as a guideline to practice decision making. A workshop was chosen rather than other methods of presenting the guideline so that participants could receive feedback and guidance from the instructors and from the other participants. Active learning educational environment will be encouraged and the workshop require group and individual participation and also assist the participants in reflection on their decisions.
  Arms: Clinical Decision Making (CDM) Workshop
Other: Clinical Decision Making (CDM) Workbook — Participants are encouraged to read and do exercises which was written in the workbook for a week and they also are asked to recall their recent patient case or use their patient as the example case and answer the questions from the Clinical Decision Making workbook.
  Arms: Clinical Decision Making Workbook

SUMMARY:
This study aims to improve the Clinical Decision Making (CDM) skills of a group of Myanmar physical therapists by series of educational workshops that will introduce them to and guide them through the decision making process by using the CDM workbook. Participants will be separated into two groups, CDM workshop group and CDM workbook group. There will be three time assessments; one pre-workshop/ workbook and two post-workshop/workbook assessments by using Clinical Decision Making (CDM) assessment worksheet.

DETAILED DESCRIPTION:
This study aims to improve the clinical decision making skills of a group of Myanmar Physical therapists by series of educational workshops that will introduce them to and guide them through the decision making process. The hypothesis of the study is the independent variable of CDM education workshop will affect the dependent variable of CDM skills of participants and the direction will be one-tailed.

Regarding my study design with pre-test-post-test for the same subjects design, samples would need 27 samples to see average change in knowledge (CDM knowledge) from pre-test to post-test with the alpha 0.05, power 0.08 and medium effect size of 0.5. However, Researcher will recruit 34 participants to cover 20% of drop out for each group. Altogether 68 participants will be needed.

Participants will be separated into two groups, one workshop and one workbook group. Among all registrants (by initial online announcement of CDM workshop and onsite invitation of CDM workshop -snow ball recruitment ), participants will be randomly assigned to two different group first then principle investigator will inform again them about their group with information sheet and informed consent form to have agreement to join the study from one group. Intervention group will have Clinical Decision Making (CDM) workshop while workbook group will be provided by the Clinical Decision Making (CDM) workbook without attending workshop and onsite interaction.

To conduct the study "Effectiveness of Clinical Decision Making (CDM) workshop in group of Myanmar Physical Therapists" , three preliminary studies have to be done before conducting the main study. Three preliminary studies are 1) Development of Clinical Decision Making (CDM) assessment worksheet, Qualitative Approach (in-depth interview) with 18 physical therapists form Yangon, 2) Validity and Reliability study of Clinical Decision Making (CDM) assessment worksheet and 3) Development of series of Clinical Decision Making (CDM) workshop based on the emerged themes and developed categories to represent the CDM knowledge in Myanmar physical therapists. Study 1 and 3 were done in order to able to develop the protocol of the main study.

Study 4: Effectiveness of Clinical Decision Making (CDM) workshop in group of Myanmar Physical Therapists

Intervention group:

* Clinical Decision Making (CDM) workshops will be presented on four weekdays and will be held in University of Medical Technology, Yangon, Myanmar in 2017.
* Participants will sign an informed consent form describing the benefits and risks of the workshops.
* Participants will be assigned a number. They will put the number on the top of the worksheet to protect their identity.
* A demographic sheet will be given during the workshop registration. This will ask participants their age, gender, years of practice, school attended, places they have practiced, area of practice specialty i.e. Pediatrics, Musculoskeletal etc.
* The workshop will begin with the first assessment approximately 30 minutes.
* During the educational workshop the CDM workbook will be presented and followed by participants as they actively sequence through a typical patient case they have chosen.
* A workbook will be used throughout the workshop which integrates the two clinical practice models: the ICF and Therapeutic Process (TP).
* The workshop will encourage and require group and individual participation and also assist the participants in reflection on their decisions.
* Participants will be assigned into small groups to introduce each other and then introduce to large group.
* Participant will choose a recent patient case and will be guided through the CDM process during the workshop using that case as their example.
* Then discussion will follow guiding the participants through the Therapeutic Process, the ICF and reflecting on choices they made or could make with the patient. During the last half hour of the last session the participants will retake the assessment worksheet.
* The CDM assessment worksheet will be administered one month at the conclusion of the workshop.
* At the time of one month post-CDM workshop assessment, participants will also be asked to reveal the number of patient cases they used CDM workbook to guide their CDM process in their practice to see usefulness of CDM workbook and opportunity to use workbook.

Workbook group:

* Participants will receive Clinical Decision Making (CDM) workbook which will be used to teach the CDM process in the four days CDM workshop.
* Participants will sign an informed consent form describing the benefits and risks of the study.
* Participants will be assigned a number. They will put the number on the top of the worksheet to protect the identity.
* Before receiving CDM workbook, participants will take the first CDM assessment it will take approximately 30 mins.
* A demographic sheet will be given before taking the first CDM assessment. This will ask participants their age, gender, years of practice, school attended, places they have practiced, area of practice specialty i.e. Pediatrics, Musculoskeletal etc.
* After one week, participants will take the second CDM assessment worksheet which is the same time with the immediate post-CDM workshop assessment of the intervention group.
* Then the CDM assessment worksheet will be administered at one month later which is the same time with the one month post-CDM workshop assessment of the intervention group.
* At the time of taking CDM assessment for the last time, participants will be asked to reveal the number of patient cases they used CDM workbook to guide their CDM process in their practice to see usefulness of CDM workbook and opportunity to use workbook.

ELIGIBILITY:
Inclusion Criteria:

* Currently practicing physical therapists with at least two years of clinical experiences.
* Participants have to be available to join all the 4 days of CDM workshop which will be held at the University of Medical Technology (UMT), Yangon, Myanmar.

Exclusion Criteria:

* Physical therapists with less than 2 years of clinical experiences.
* Physical therapists who were not educated in Myanmar.
* Physical therapists who are not available to join all 4 days of CDM workshop.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
Pre-Intervention Clinical Decision Making (CDM) Assessment | Baseline (before intervention)
  The CDM worksheet represents the knowledge for four main elements of Clinical Decision Making (CDM) process; Health Condition, Examination, Evaluation and Intervention. These four elements represent the sequence of content which will include in the CDM education workshop. The CDM Assessment Worksheet includes three types of question: two categorical measurement level and one open-ended qualitative type of question.
Immediate-post Intervention Clinical Decision Making (CDM) Assessment | Immediate post-Intervention
  The CDM worksheet represents the knowledge for four main elements of Clinical Decision Making (CDM) process; Health Condition, Examination, Evaluation and Intervention. These four elements represent the sequence of content which will include in the CDM education workshop. The CDM Assessment Worksheet includes three types of question: two categorical measurement level and one open-ended qualitative type of question.
One month post-Intervention Clinical Decision Making (CDM) Assessment | One-month post-Intervention
  The CDM worksheet represents the knowledge for four main elements of Clinical Decision Making (CDM) process; Health Condition, Examination, Evaluation and Intervention. These four elements represent the sequence of content which will include in the CDM education workshop. The CDM Assessment Worksheet includes three types of question: two categorical measurement level and one open-ended qualitative type of question.

CONTACTS AND LOCATIONS:
Overall Officials: Phyu H Hlaing, PhD, Principal Investigator — Mahidol University
Locations (1):
- University of Medical Technology, Yangon, Insein, Burma

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wainwright SF, Shepard KF, Harman LB, Stephens J. Factors that influence the clinical decision making of novice and experienced physical therapists. Phys Ther. 2011 Jan;91(1):87-101. doi: 10.2522/ptj.20100161. Epub 2010 Dec 2. PMID 21127167
- [Background] Wainwright SF, Shepard KF, Harman LB, Stephens J. Novice and experienced physical therapist clinicians: a comparison of how reflection is used to inform the clinical decision-making process. Phys Ther. 2010 Jan;90(1):75-88. doi: 10.2522/ptj.20090077. Epub 2009 Nov 19. PMID 19926680